CLINICAL TRIAL: NCT05444010
Title: Mandala Intervention on Mental Health Problems of Nurses Caring for Terminally Ill Patients
Brief Title: Mandala Intervention on Mental Distress in Nurses Working With Terminally Ill Patients
Acronym: mandala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Arzu Nurdaş, Principal investigator, Istanbul Sabahattin Zaim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISZU
Record Dates: First submitted 2022-06-16; First posted 2022-07-05 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Mental Health Issue
Keywords: mental health, anxiety, depression
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control grups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mental health (Experimental): The effect of mandala painting on mental health. Mental health-related anxiety, depression, well-being, distress and death anxiety and depression will be measured.
  Interventions: Behavioral: mandala painting

INTERVENTIONS:
Behavioral: mandala painting — nurse painted mandala for relaksing

SUMMARY:
Mandala application intervention of mental distress in nurses working with terminally ill patients

DETAILED DESCRIPTION:
Questionnaires were applied to the control and experimental groups. Mandala painting was done to the experimental group. Questionnaires were applied to the control and experimental groups again. Distress, anxiety, depression, death anxiety, death depression and psychological well-being of the experimental and control groups were evaluated.

ELIGIBILITY:
Inclusion Criteria:

volunteer

* active employee
* year of study

Exclusion Criteria:

* paint allergy
* use of psychiatric drugs Loss of loved one in the last six months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Beck depresion scale | 4 week
  depresion is mental breakdown, depresion for beck depresion scale, 0-9 depresion emity, 10-15 light depression, 16-23 middle depresion, 24- 63 severe depression

SECONDARY OUTCOMES:
STAI-trait anxiety scale | 4 week
  anxiete is boredom, anxiete for trait anxiety scale, 0-15 anxiety none,n , 15-30 light anxiety, 30-60 middle anxiety, over 60 severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: RUKİYE PINAR BÖLÜKTAŞ, Study Director — SZU
Locations (2):
- Turkey (Türkiye) (2):
  - SZU, Istanbul, İSTANBUL/halkalı
  - SZU, Istanbul, İ̇stanbul

IPD SHARING:
Plan to Share IPD: Yes
mandala painting 4 week
Supporting Information: Study Protocol, SAP
Time Frame: mayıs 2022-haziran 2022
Access Criteria: emity